CLINICAL TRIAL: NCT00453349
Title: A Prospective, Randomized, Double Dummy, Double Blind, Multi-center Multinational Trial Comparing the Efficacy and Safety of Moxifloxacin 400 mg PO QD 24 Hours for 14 Days to That of Levofloxacin 500 mg PO QD 24 Hours Plus Metronidazole 500 mg BID for 14 Days in Subjects With an Uncomplicated Pelvic Inflammatory Disease (PID). Moxifloxacin, Metronidazole, and Levofloxacin in Asia (MONALISA Study)
Brief Title: A Trial Comparing Moxifloxacin Versus Levofloxacin Plus Metronidazole In Uncomplicated Pelvic Inflammatory Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11981; 2006-000874-56 (EudraCT Number)
Record Dates: First submitted 2007-03-27; First posted 2007-03-28 (Estimated); Results first posted 2009-11-30 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-09

CONDITIONS: Pelvic Inflammatory Disease
Keywords: Uncomplicated pelvic inflammatory disease
MeSH Terms: conditions — Pelvic Inflammatory Disease | interventions — Moxifloxacin; Levofloxacin; Metronidazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moxifloxacin (Experimental): Moxifloxacin (Avelox, BAY12-8039) 400 mg by mouth (PO) once daily for 14 days
  Interventions: Drug: Moxifloxacin (Avelox, BAY12-8039)
- Levofloxacin plus Metronidazole (Active Comparator): Levofloxacin 500 mg by mouth (PO) once daily for 14 days plus Metronidazole 500 mg (PO) twice daily for 14 days
  Interventions: Drug: Levofloxacin & Metronidazole

INTERVENTIONS:
Drug: Moxifloxacin (Avelox, BAY12-8039) — Moxifloxacin (Avelox, BAY12-8039) 400 mg by mouth (PO) once daily for 14 days
  Arms: Moxifloxacin
Drug: Levofloxacin & Metronidazole — Levofloxacin 500 mg by mouth (PO) once daily for 14 days plus Metronidazole 500 mg (PO) twice daily for 14 days
  Arms: Levofloxacin plus Metronidazole

SUMMARY:
To assess the efficacy and safety of oral moxifloxacin compared to oral levofloxacin plus oral metronidazole in uncomplicated pelvic inflammatory disease (PID)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of uncomplicated PID based on the absence of pelvic or tubo-ovarian abscess at pelvic ultrasound and/or laparoscopic examination.

Exclusion Criteria:

* Subjects with impaired liver and renal function; known hypersensitivity to study drugs, related compounds or any of the excipients.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2007-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (12):
- China (5):
  - Shenyang, Liaoning
  - Chengdu, Sichuan
  - Beijing
  - Chongqing
  - Shanghai
- Jakarta, Indonesia
- Karachi, Pakistan
- Manila, Philippines
- Seoul, South Korea
- Taiwan (2):
  - Taipei, Taiwan
  - Taizung
- Bangkok, Bangkok, Thailand

REFERENCES:
- [Result] Judlin P, Liao Q, Liu Z, Reimnitz P, Hampel B, Arvis P. Efficacy and safety of moxifloxacin in uncomplicated pelvic inflammatory disease: the MONALISA study. BJOG. 2010 Nov;117(12):1475-84. doi: 10.1111/j.1471-0528.2010.02687.x. Epub 2010 Aug 18. PMID 20716255

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 463 females with uncomplicated PID were enrolled on the basis of a complete evaluation (interview, medical history and physical examination and laboratory tests). 460 subjects were randomized, 412 completed study treatment (whole medication), and 384 subjects were valid for the primary efficacy analysis.
Pre-assignment Details: The efficacy results in ITT are consistent with those in PP, supporting that this is a non-inferiority study and the primary efficacy population was PP not ITT. 76 subjects were excluded from primary efficacy analysis mainly due to essential data missing or invalid, violation of inclusion/exclusion criteria and insufficient duration of therapy.
Period: Randomized
Arm/Group | Moxifloxacin | Levofloxacin Plus Metronidazole
Started | 228 | 232
Completed | 203 | 209
Not Completed | 25 | 23
Not completed — Adverse Event | 12 | 11
Not completed — Lack of Efficacy | 2 | 1
Not completed — Lost to Follow-up | 7 | 5
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 3 | 5
Period: Reaching of Primary Endpoint (TOC)
Arm/Group | Moxifloxacin | Levofloxacin Plus Metronidazole
Started | 225 (Subjects who attended the TOC visit or at least had a clinical evaluation at TOC) | 230 (i.e. the ITT population)
Valid for Primary Efficacy Analysis | 194 | 190
Completed | 215 (All PP patients and ITT patients with a clinical response with no missing information) | 219
Not Completed | 10 | 11
Not completed — Missing information | 10 | 11
Period: Completed Study
Arm/Group | Moxifloxacin | Levofloxacin Plus Metronidazole
Started | 228 | 232
Completed Study Treatment | 203 (25 terminated prematurely) | 209 (23 terminated prematurely)
Completed | 201 (had follow-up assessment or alternative antibiotic assessment) | 198 (had follow-up assessment or alternative antibiotic assessment)
Not Completed | 27 | 34
Not completed — Adverse Event | 12 | 11
Not completed — Lack of Efficacy | 2 | 1
Not completed — Lost to Follow-up | 7 | 5
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 3 | 5
Not completed — Lost to follow up after study treatment | 2 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moxifloxacin | Levofloxacin Plus Metronidazole | Total
Number analyzed (Participants) | 228 | 232 | 460
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.2 (8.4) | 35.4 (8.7) | 35.2 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 228 | 232 | 460
  Male | 0 | 0 | 0
Microbiology recovery [Number; unit: number of participants with pathogenes] — Endocervical samples were taken for culture and Polymerase Chain Reaction (PCR) tests within 48 hours prior to start of therapy. The PCR tests were repeated at TOC and Follow-up visits if the pre-therapy results were positive for Neisseria gonorrhoeae and Chlamydia trachomatis.
  number of participants with pathogenes | 36 | 36 | 72
Total pelvic pain score (using modified McCormack score) [Mean (Standard Deviation); unit: points on a scale] — Modified McCormack score was used to assess the tenderness at the abdominal and pelvic examination, 0=tenderness absent, 1=tenderness described by the subject but not manifested by facial expression or muscle tone changes, 2=tenderness resulting in altered facial expression or muscle tone, 3=tenderness causing observable marked distress.
  points on a scale | 11.3 (3.8) | 11.6 (3.8) | 11.5 (3.8)

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response 7 to 14 Days After Completion of Study Drug Therapy in Per Protocol (PP) Population
Description: Clinical cure was defined as: Reduction of the tenderness score (modified McCormack) by > 70% and apyrexia (rectal/tympanic/oral temperature value < 38.0°C or axillary temperature value < 37.5°C) and white blood cell count < 10,500/mm^3.
Time Frame: 7 - 14 days after completion of study drug therapy
Population: The number of subjects in the PP population was slightly higher than the planned number of subjects (184 subjects per treatment group). The most common reasons for exclusion from the population valid for efficacy in both the Moxifloxacin and Comparator were essential data missing/invalid, followed by violation of inclusion/exclusion criteria.
Measure: Number; unit: participants
Arm/Group | Moxifloxacin | Levofloxacin Plus Metronidazole
Number analyzed (Participants) | 194 | 190
participants
  Clinical cure | 152 | 155
  Clinical non-success | 42 | 35
Statistical Analysis 1: Comparison: Moxifloxacin vs Levofloxacin Plus Metronidazole; Calculated were 95% confidence intervals for the difference in success rates between treatment groups (moxifloxacin minus comparator). Method as described in Koch et al. ('Categorical Data Analysis' in Statistical methodology in the pharmaceutical sciences / edited by D. A. Berry, p. 415 ff., Marcel Dekker, 1990); Test type: Non-Inferiority or Equivalence — The non-inferiority margin was set to 15% in the protocol. Sample size was estimated using the method as described in Farrington-Manning (STATISTICS IN MEDICINE, Vol. 9; Farrington CP, Manning G: "Test statistics and sample size formulae for comparative binomial trials with null hypothesis of non-zero risk difference...", pg.1447-1454 [1990]). Estimation was performed to achieve 90% power, based on the equivalence delta of 15%, and a clinical success rate of 87% in the per protocol population; Mean Difference (Final Values) = -3.2, 95% CI [-10.7 to 4.9] — Mean difference denotes the difference of clinical cure rates in percent between the two treatment groups. A positive value indicates an advantage for the treatment group of moxifloxacin, a negative value an advantage for the comparator group

2. Secondary Outcome: Clinical Response 7 to 14 Days After Completion of Study Drug Therapy on Intent To Treat (ITT) Population
Description: For any subject in the ITT population also valid for the PP analysis, same clinical response as in the PP analysis was applied to the ITT analysis. For those subjects in the ITT population invalid for the PP analysis, any clinical response different from clinical cure was set to "non-success".
Time Frame: 7 - 14 days after completion of study drug therapy
Population: Subjects who were randomized, had received at least one dose of study medication and had at least one observation after drug intake would be included in the ITT analysis.
Measure: Number; unit: participants
Arm/Group | Moxifloxacin | Levofloxacin Plus Metronidazole
Number analyzed (Participants) | 225 | 230
participants
  Clinical cure | 163 | 171
  Clinical non-success | 62 | 59
Statistical Analysis 1: Comparison: Moxifloxacin vs Levofloxacin Plus Metronidazole; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Sample size estimation was based on the primary efficacy variables; Mean Difference (Final Values) = -1.9, 95% CI [-9.9 to 6.0] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Clinical Response on Treatment for Per Protocol Population
Description: At the During Therapy (Day 4 to 7) assessment, the clinical response was graded as clinical Improvement (severity score reduced by >30% with improvement in temperature, clinical failure (reduction in severity score of < or equal 30% and/or no improvement in temperature) or indeterminate (clinical assessment not possible to determine).
Time Frame: 4 - 7 days after start of therapy
Population: Analysis was performed for the per protocol population.
Measure: Number; unit: participants
Arm/Group | Moxifloxacin | Levofloxacin Plus Metronidazole
Number analyzed (Participants) | 188 | 186
participants
  Clinical Improvement | 177 | 181
  Clinical failure | 11 | 5
Statistical Analysis 1: Comparison: Moxifloxacin vs Levofloxacin Plus Metronidazole; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Sample size estimation was based on the primary efficacy variables; Mean Difference (Final Values) = -3.2, 95% CI [-7.4 to 0.8] — Mean difference denotes the difference of clinical improvement rates in percent between the two treatment groups. A positive value indicates an advantage for the treatment group of moxifloxacin, a negative value an advantage for the comparator group

4. Secondary Outcome: Clinical Response on Treatment for Intent To Treat Population
Description: Clinical response during treatment was analyzed exploratively in the same way as the primary efficacy variable. At the During Therapy (Day 4 to 7) assessment, the clinical response was graded as clinical Improvement, clinical failure or indeterminate accordingly. Clinical improvement was considered success, all other outcomes as non-success.
Time Frame: 4 - 7 days after start of therapy
Population: Subjects who were randomized, had received at least one dose of study medication and had at least one observation after drug intake would be included in the ITT analysis. For any subject in the ITT population also valid for the PP analysis, same clinical response as in the PP analysis was applied to the ITT analysis.
Measure: Number; unit: participants
Arm/Group | Moxifloxacin | Levofloxacin Plus Metronidazole
Number analyzed (Participants) | 225 | 230
participants
  Clinical improvement | 166 | 170
  Failure, indeterminate, missing | 59 | 60
Statistical Analysis 1: Comparison: Moxifloxacin vs Levofloxacin Plus Metronidazole; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Sample size estimation was based on the primary efficacy variables; Mean Difference (Final Values) = -0.1, 95% CI [-8.1 to 7.5] — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: Bacteriological Response at Test Of Cure (TOC) Visit Microbiologically Valid
Description: The bacteriological responses was based on the results of appropriate cultures taken before and, if necessary, during treatment, at the TOC visit and within the follow-up period. Bacteriological response at the TOC visit would also be based on repeated PCR tests for N. gonorrhoeae and C. trachomatis.
Time Frame: 7 - 14 days at TOC visit
Population: All subjects for whom a specific bacterial pathogen was isolated/identified from any pre-treatment culture and which was considered responsible for the infection would be assessed for bacteriological efficacy.
Measure: Number; unit: participants
Arm/Group | Moxifloxacin | Levofloxacin Plus Metronidazole
Number analyzed (Participants) | 30 | 26
participants
  Eradication | 27 | 22
  Persistence | 3 | 4
Statistical Analysis 1: Comparison: Moxifloxacin vs Levofloxacin Plus Metronidazole; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Sample size estimation was based on the primary efficacy variables; Mean Difference (Final Values) = 5.4, 95% CI [-12.7 to 20.3] — Mean difference denotes the difference of eradication rates in percent between the two treatment groups. A positive value indicates an advantage for the treatment group of moxifloxacin, a negative value an advantage for the comparator group

6. Secondary Outcome: Bacteriological Response at Test Of Cure (TOC) Visit in Intent To Treat Population With Causative Organism
Description: Bacteriological response at the TOC was analyzed exploratively in the same way as the primary efficacy variable based on the subgroup of microbiologically valid subjects. At the TOC visit, eradication was considered a bacteriological success, and persistence, presumed persistence and superinfection were considered bacteriological failures.
Time Frame: 7 - 14 days at TOC visit
Population: Patients were included in this analysis if a causative organism could be established pre-therapy by culture or PCR, and if the patient was valid for intent-to-treat.
Measure: Number; unit: participants
Arm/Group | Moxifloxacin | Levofloxacin Plus Metronidazole
Number analyzed (Participants) | 36 | 34
participants
  Eradication | 28 | 25
  Persistence, indeterminate, missing | 8 | 9
Statistical Analysis 1: Comparison: Moxifloxacin vs Levofloxacin Plus Metronidazole; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Sample size estimation was based on the primary efficacy variables; Mean Difference (Final Values) = 4.3, 95% CI [-19.4 to 17.6] — [estimate comment as in outcome 5, analysis 1]

7. Secondary Outcome: Clinical Response at Follow-up Visit on Per Protocol Population
Description: Clinical response at follow up was analyzed exploratively in the same way as the primary efficacy variable. At Follow-up, the clinical response was graded as continued cure, clinical relapse, or indeterminate, of which only continued cure was considered success. Failures from end of treatment were carried forward.
Time Frame: 28 - 42 days after completion of study drug therapy
Population: All successfully treated subjects and subjects evaluated as "indeterminate" at TOC, who were not administered an additional antibiotic therapy would have their clinical response rate assessed at the follow up visit. Patients with missing or indeterminate outcome were omitted.
Measure: Number; unit: participants
Arm/Group | Moxifloxacin | Levofloxacin Plus Metronidazole
Number analyzed (Participants) | 184 | 180
participants
  Continued clinical cure | 157 | 158
  Continued failure, clinical recurrence/relapse | 27 | 22
Statistical Analysis 1: Comparison: Moxifloxacin vs Levofloxacin Plus Metronidazole; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Sample size estimation was based on the primary efficacy variables; Mean Difference (Final Values) = -2.5, 95% CI [-8.6 to 4.9] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Clinical Response at Follow-up Visit on Intent To Treat Population
Description: All successfully treated subjects and subjects evaluated as"indeterminate" at TOC, who were not administered an additional antibiotic therapy would have their clinical response rate assessed at the follow-up visit. Patients with missing or indeterminate outcome were treated as non-successes.
Time Frame: 28 - 42 days after completion of study drug therapy
Population: At the follow-up visit, the clinical response in subjects who were non-failures at the TOC visit were graded as Continued cure, Clinical relapse or Indeterminate.
Measure: Number; unit: participants
Arm/Group | Moxifloxacin | Levofloxacin Plus Metronidazole
Number analyzed (Participants) | 225 | 230
participants
  Continued clinical cure | 166 | 170
  Failure, relapse, indeterminate, missing | 59 | 60
Statistical Analysis 1: Comparison: Moxifloxacin vs Levofloxacin Plus Metronidazole; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Sample size estimation was based on the primary efficacy variables; Mean Difference (Final Values) = -0.1, 95% CI [-8.1 to 7.5] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Bacteriological Response at Follow-up Visit Microbiologically Valid
Description: Subjects with at least one causative organism identified in the pre-therapy culture or a positive pre-therapy PCR result and an appropriate post-therapy bacteriological evaluation available were analyzed. Bacteriological responses at follow-up visit was analyzed exploratively in the same way as the primary efficacy variable.
Time Frame: 28 - 42 days after completion of study drug therapy
Population: At the follow-up visit, the bacteriological success response was classified as eradication, and recurrence/persistence as bacteriological failures.
Measure: Number; unit: participants
Arm/Group | Moxifloxacin | Levofloxacin Plus Metronidazole
Number analyzed (Participants) | 28 | 26
participants
  Eradication | 23 | 22
  Eradication with recurrence, persistence | 5 | 4
Statistical Analysis 1: Comparison: Moxifloxacin vs Levofloxacin Plus Metronidazole; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Sample size estimation was based on the primary efficacy variables; Mean Difference (Final Values) = -7.9, 95% CI [-24.9 to 15.9] — [estimate comment as in outcome 5, analysis 1]

10. Secondary Outcome: Bacteriological Response at Follow-up Visit in Intent To Treat Population With Causative Organism
Description: as for outcome 9
Time Frame: 28 - 42 days after completion of study drug therapy
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | Moxifloxacin | Levofloxacin Plus Metronidazole
Number analyzed (Participants) | 36 | 34
participants
  Eradication | 23 | 23
  Eradication with recurrence, persistence | 13 | 11
Statistical Analysis 1: Comparison: Moxifloxacin vs Levofloxacin Plus Metronidazole; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Sample size estimation was based on the primary efficacy variables; Mean Difference (Final Values) = 3.7, 95% CI [-30.5 to 11.9] — [estimate comment as in outcome 5, analysis 1]

11. Secondary Outcome: Number of Subjects Who Received Alternative Medicine
Description: As alternative medicine any systemic antibacterial medication was considered.
Time Frame: Up to 42 days after end of treatment
Population: The number of subjects who received alternative medicine in the PP population was analyzed. The clinical response was graded as alternative medicine (clinical cure, improvement, continued clinical cure) versus no alternative medicine.
Measure: Number; unit: participants
Arm/Group | Moxifloxacin | Levofloxacin Plus Metronidazole
Number analyzed (Participants) | 194 | 190
participants
  Receiving alternative medicine | 4 | 1
  Not receiving alternative medicine | 190 | 189

ADVERSE EVENTS:
Arm/Group | Moxifloxacin | Levofloxacin Plus Metronidazole
Serious Adverse Events (participants affected / at risk) | 3/225 | 1/230
Other Adverse Events (participants affected / at risk) | 83/225 | 94/230
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Moxifloxacin (N=225) | Levofloxacin Plus Metronidazole (N=230)
Colitis (Gastrointestinal disorders) | 1 | 0
Pyelonephrits acute (Infections and infestations) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Moxifloxacin (N=225) | Levofloxacin Plus Metronidazole (N=230)
Abdominal pain upper (Gastrointestinal disorders) | 10 | 14
Nausea (Gastrointestinal disorders) | 43 | 54
Vomiting (Gastrointestinal disorders) | 7 | 15
Dizziness (Nervous system disorders) | 39 | 36
Insomnia (Psychiatric disorders) | 7 | 14

LIMITATIONS AND CAVEATS:
Out of the 460 randomized subjects, 5 subjects (3 moxifloxacin subjects, 2 placebo subjects) did not receive any study medication. Only one of these patients had an adverse event (stomachache, randomized to Moxifloxacin).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less